CLINICAL TRIAL: NCT05000229
Title: Residual Symptoms in Patients With a History of Coronavirus Disease (COVID-19) and Their Impact on Biopsychosocial Functions (Post-Covid Syndrome)
Brief Title: Residual Symptoms After Coronavirus Disease (COVID-19) in Lithuanian Population
Acronym: Post-Covid
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lithuanian University of Health Sciences (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Dovilė Važgėlienė, MD, PhD-student, Lithuanian University of Health Sciences
Other Study IDs: 001/Version 1
Record Dates: First submitted 2021-07-16; First posted 2021-08-11 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Post-Covid Syndrome
Keywords: Post-Covid syndrome; Rehabilitation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to describe the post-covid-19 syndrome in Lithuanian population regarding the remaining symptoms and their impact on physical functioning, work ability and needs of rehabilitation.

DETAILED DESCRIPTION:
Participants with suspected and confirmed cases of COVID-19 infection will complete an anonymous online questionnaire for post-covid syndrome, i.e. symptoms lasting longer than 28 days after post-covid-19 syndrome. The online survey is developed to assess the health state before infection and residual symptoms lasting longer than acute COVID-19 infection, influencing the functional activity and work ability. The needs of rehabilitation will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years age patients;
* a history of COVID-19 infection that was and was not positive for SARS-CoV-2 diagnostic or antibody testing
* the duration of remaining symptoms is longer than 28 days
* ability to fulfil internet-based questionnaire

Exclusion Criteria:

* ongoing covid-19 infection
* other comorbidities requiring treatment or rehabilitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The online study will be open to all volunteers over the age of 18 with COVID-19 infection
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-05-04 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Description of post-covid-19 syndrome in Lithuanian population | 2021.05.04 - 2022.12.31
  Post-covid-19 syndrome in Lithuanian population: prevalence, symptomatology and needs of rehabilitation

SECONDARY OUTCOMES:
Assessment of medical premorbid status in post-covid-19 syndrome | 2021.05.04 - 2022.12.31
  The severity of comorbidities in terms of self-reported medical diagnoses and medication

CONTACTS AND LOCATIONS:
Locations (1):
- Lithuanian University of Health Sciences, Kaunas, Lithuania